CLINICAL TRIAL: NCT06015659
Title: Phase 2 Single Arm Trial Testing the ZN-c3 WEE1 Inhibitor in Combination With Gemcitabine in Second-Line Advanced Pancreatic Adenocarcinoma
Brief Title: ZN-c3 + Gemcitabine in Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brandon Huffman, MD (Other)
Collaborators: Lustgarten Foundation (Other); K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor-Investigator, Brandon Huffman, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-336
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Advanced Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZN-c3 + Gemcitabine (Experimental): Study procedures will be conducted as follows:
  * Cycle 1 - End of Treatment
    * Days 1 - 5 of 21-day cycle: Predetermined dose of ZN-c3 1x daily.
    * Days 8 - 12 of 21-day cycle: Predetermined dose of ZN-c3 1x daily.
    * Days 15 - 19 of 21-day cycle: Predetermined dose of ZN-c3 1x daily.
    * Day 1 and 8 of 21-day cycle: Predetermined dose of Gemcitabine 1x daily.
  * On-treatment tumor biopsy will be collected on either Cycle 1 Day 9 - 10 or Cycle 2 Day 9 - 10.
  * Tumor assessment by Computerized Tomography (CT) or Magnetic Resonance Imaging scan every 8 weeks while on treatment.
  * End of treatment visit with tumor assessment by CT or MRI and optional tumor biopsy.
  * Follow up visit every 2 months after treatment has ended.
  Interventions: Drug: Zentalis; Drug: Gemzar

INTERVENTIONS:
Drug: Zentalis — Small molecule inhibitor of the WEE1 tyrosine kinase, tablet taken orally per protocol.
  Other Names: Zn-c3, KP-2638, azenosertib, C29H34N8O2.
Drug: Gemzar — Nucleoside metabolic inhibitor, per standard care via intravenous infusion.
  Other Names: Gemcitabine hydrochloride, FF 10832, LY188011, C9H11F2N3O4 - HCl

SUMMARY:
This study is being done to test the safety and effectiveness of combining ZN-c3 and Gemcitabine in participants with pancreatic cancer.

The names of the study drugs involved in this study are:

* ZN-c3 (a small molecule inhibitor of the WEE1 tyrosine kinase)
* Gemcitabine (a nucleoside metabolic inhibitor)

DETAILED DESCRIPTION:
This is an open label, single arm phase 2 trial evaluating ZN-c3 combined with gemcitabine in second-line advanced pancreatic cancer. There are lab experiments that show that pancreatic cancer cells can respond to a combination of ZN-c3, an experimental drug, with gemcitabine.

The U.S. Food and Drug Administration (FDA) has not approved ZN-c3 as a treatment for any disease. The FDA has approved gemcitabine as a treatment option for advanced pancreatic cancer.

The research study procedures include screening for eligibility, study treatment including evaluations and follow up visits, radiological scans (Computerized Tomography, Magnetic Resonance Imaging, or Positron Emission Tomography), blood tests, electrocardiogram, and tumor biopsy.

It is expected that about 34 people will take part in this research study.

The Lustgarten Foundation for Pancreatic Research and Stand Up to Cancer are supporting this research study by providing funding to conduct the study. Zentalis is supplying the study drug, ZN-c3.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pathologically confirmed advanced pancreatic adenocarcinoma that is not curable with standard approaches based on the judgement of the treating investigator. Patients with metastatic pancreatic cancer and unresectable pancreatic cancer are eligible.
* Patients must have progressed or not tolerated a platinum-based regimen prior to enrolling on the trial.
* Patients must have received no more than 1 prior lines of platinum-based chemotherapy in the metastatic setting. Therapy given in the adjuvant or neoadjuvant setting is counted as a prior therapy if it occurred less than 6 months before cancer recurrence or progression.
* Age ≥ 18 years. As no dosing or adverse event data are currently available in participants < 18 years of age, children and adolescents are excluded from this study.
* ECOG performance status of 0 or 1 (see Appendix A) with no deterioration over the previous 2 weeks prior to day of first dosing (Cycle 1, Day 1).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3 excluding measurements obtained within 3 days after transfusion of platelets
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN); or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with documented Gilbert's Syndrome.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) Albumin ≤2.5 x institutional ULN; ≤ 5 × institutional ULN if liver metastases ≥ 2.7 g/dL
  * Creatinine clearance (CrCl) ≥ 50 ml/min based on Cockroft-Gault method
* Participants must have measurable disease by RECIST v. 1.1 criteria and be willing to undergo a pre-treatment and on-treatment tumor biopsy. The biopsy requirement can be waived only with approval from the sponsor-investigator.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated, unless there is a drug-drug interaction with study medication.
* Patient has read and understands the informed consent form (ICF) and has been given written ICF prior to any study procedures which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Female patients who are not of child-bearing potential* and women of childbearing potential who agree to use adequate contraceptive measures prior to the first dose and for 90 days after the last dose of ZN-c3, and who have a negative serum or urine pregnancy test within 14 days prior to the start of study treatment.

  --Evidence of non-childbearing status, defined as below:
  * Women who are surgically sterile (i.e., have undergone bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy).
  * Age ≥50 years with any one or more of the conditions below:

    * Amenorrheic for 12 months or more following cessation of all hormonal replacement therapy
    * Had radiation-induced menopause with last menses >1 year ago
    * Had chemotherapy-induced menopause with last menses >1 year ago
  * Age <50 if amenorrhoeic for 12 months or more following cessation of all hormonal replacement therapy and if luteinizing hormone and follicle- stimulating hormone levels are in the post-menopausal range per institutional standards of practice.
* Male patients should be willing to abstain or use barrier contraception (i.e., condoms) for the duration of the study drug exposure and for 90 days after the last dose of ZN- c3 after study treatment discontinuation.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load, unless there is a drug-drug interaction with study medication.

Exclusion Criteria:

* Patients who have previously received a WEE1 inhibitor are not eligible.
* Patients who received gemcitabine for incurable pancreatic cancer (locally advanced unresectable or metastatic) or patients progressing within 6 months of receiving neoadjuvant/adjuvant gemcitabine.
* Use of an anti-cancer treatment drug ≤ 21 days or 5 half-lives (whichever is shorter) prior to the first dose of ZN-c3.
* Active use of treatment prescription or non-prescription drugs, or food and herbal supplements, that are strong/moderate CYP3A4 inhibitors, P-gp inhibitors, or strong CYP3A4 inducers.
* Any prior palliative radiation to ≥5% of the bone marrow, and must have been completed and recovered from adverse effects of therapy at least 21 days prior to the first dose of ZN-c3.
* Participants who have undergone major surgical procedures ≤ 28 days, or minor surgical procedures ≤ 7 days, of the first dose of ZN-c3. No waiting period is required following port-a-cath or other central venous access placement.
* Presence of CTCAE v5.0 Grade >1 toxicity from prior therapy (except alopecia, anorexia or CTCAE grade 2 peripheral neuropathy).
* Patient is unable to swallow oral medications. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN).
* Participants with known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or hemorrhage for at least 2 weeks after the completion of treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrollment.
* History of hypersensitivity to compounds of similar chemical or biologic composition to gemcitabine or ZN-c3.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection*, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements.
* Recurrent, active or suspected infection and/or patients who are predisposed to an increased risk of severe infection. Patients with infections that require antibiotics or antifungal agents may be eligible, provided that infection is resolved and treatment is completed at least 7 days prior to study treatment start.
* Participants with a clinically significant gastrointestinal disorder that in the opinion of the treating investigator could impact the absorption of the study drugs, including but not limited to refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of ZN-c3.
* Participants with a history of a clinically relevant second primary malignancy within the past 2 years. Exceptions include: resected basal and squamous cell carcinomas of the skin and completely resected carcinoma in situ of any type.
* Administration of strong or moderate CYP3A4 inhibitors or inducers and P-gp inhibitors. (See Appendix B)
* Pregnant or lactating women are excluded from this study because gemcitabine/ZN- c3 are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with gemcitabine/ZN-c3, breastfeeding should be discontinued if the mother is treated with gemcitabine/ZN-c3.
* Any of the following cardiac diseases currently or within 6 months of the first dose of ZN-c3:

  * 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of >470 ms, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-Free Survival (PFS) Rate | 18 months
  6-month PFS rate is the proportion of participants remaining alive and progression free at 6 months. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | 18 months
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Median Progression-Free Survival (PFS) | 18 months
  Progression-free survival based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Objective Response Rate (ORR) | 18 months
  The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECISTv1.1 criteria.
Grade 3-5 Treatment-related Toxicity Rate | 18 months
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Huffman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu